CLINICAL TRIAL: NCT02594293
Title: A Prospective, Randomized, Controlled Clinical Trial to Evaluate the Role of Peg-IFN Alfa-2a in Reducing RelapSe Rate in Patients With Hepatitis B e Antigen(HBeAg)-nEgative Chronic Hepatitis B After Discontinuation of NUC Therapy
Brief Title: Pegylated Interferon(Peg-IFN) in Reducing Relapse Rate in Patients After Discontinuation of NUC Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Jiming Zhang, chief physician,professor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CEASE
Record Dates: First submitted 2015-10-11; First posted 2015-11-03 (Estimated); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Controlled Group (No Intervention): Discontinue the NA treatment and follow up for 96 weeks
- Pegasys 48 weeks (Experimental): Discontinue the NA treatment ,PegIFN alfa-2a 180 μg by week for 48 weeks and follow up for 48 weeks
  Interventions: Drug: PegIFN alfa-2a

INTERVENTIONS:
Drug: PegIFN alfa-2a — 180 μg/ 0.5 ml ,hypodermic injection once a week
  Other Names: Pegasys
  Arms: Pegasys 48 weeks

SUMMARY:
This study evaluates whether Peg-IFN alfa-2a can reduce the recurrence rate of hepatitis B in 96 weeks after nucleoside analogue (NUC) withdrawal.

The HBV HBeAg-Negative patients who received NUC anti-virus treatment for 2.5 years and reached stopping rule in 《Chinese chronic hepatitis B prevention and treatment guidelines》(2010) were randomly assigned into three groups: One group discontinue the NUC treatment and follow up for 96 weeks,One discontinue the NUC treatment ,receive Peg-IFN alfa-2a 180 μg by week for 24 weeks and follow up for 72 weeks,The other discontinue the NUC treatment ,receive Peg-IFN alfa-2a 180 μg by week for 48 weeks and follow up for 48 weeks.

DETAILED DESCRIPTION:
NUC is a potent inhibitor of hepatitis B viral(HBV) replication, but long-term therapy may be required. Therefore, NUC resistance is an important clinical risk resulting from long-term therapy in chronic hepatitis B (CHB) management. Discontinuation of NUC is a feasible strategy to reduce resistance. However, the high rate of relapse after cessation of NUC treatment in CHB patients remains a big problem. NUC treatment of how to safely stop drug needs to be solved.

Peg-IFN can clear HBV by direct anti-viral and immune regulation mechanisms including enhancing natural killer cell response, increased cluster of differentiation 8(CD8 +) T lymphocytes and other mechanisms to restore and enhance the immune response in patients with CHB. Response to PEG-IFN is frequently sustained after a finite treatment course due to its immune modulating capacity.

ELIGIBILITY:
Inclusion Criteria:

1. HBeAg-Negative Chronic Hepatitis B Patients：HBsAg-Positive,HBsAb-Negative,HBeAg-Negative,HBeAb-Positive during screening period and before NA treatment
2. NUC monotherapy (including adefovir and entecavir) for more than 2.5 years,and reached stopping rule in 《Chinese chronic hepatitis B prevention and treatment guidelines》(2010):the patients who achieved undetectable HBV DNA (<300 copies/mL) with normal alanine aminotransferase (ALT) and the consolidation therapy reached 1.5 years ,total course of the treatment reached 2.5 years can stop NUC therapy
3. Willing to stop the drug, and signed a written informed consent

Exclusion Criteria:

1. HBsAb positive in screening period
2. Compensated or Decompensated liver cirrhosis:with history of cirrhosis before NUC treatment or Child-Pugh score ≥ 5 or Complications of liver cirrhosis such as ascites, hepatic encephalopathy, esophageal gastric varices bleeding
3. Hypersensitivity to interferon(IFN) or its active substance, and ineligible to IFN
4. A history of immunoregulation drug therapy within one year before entry including IFN and so on.
5. Coinfection with HAV、HCV、HDV、HEV 、HIV or with Other chronic liver diseases such as Alcoholic Liver Disease,Inherited Metabolic Liver Disease,Drug induced Liver Disease and nonalcoholic fatty liver
6. Autoimmune disease including Autoimmune hepatitis and Psoriasis and so on.
7. Hepatocellular carcinoma(HCC) or alpha feto protein(AFP) levels more than 100 ng/ml and Hepatic malignant potential of Imaging examination or AFP levels more than 100 ng/ml for 3 months
8. A neutrophil count of less than 1500 per cubic millimeter or a platelet count of less than 90,000 per cubic millimeter
9. A serum creatinine level that was more than 1.5 times the upper limit of the normal range
10. With other malignant tumors(exclude the cured ones)
11. Severe organ dysfunction
12. With severe psychiatric condition or nervous disease such as epilepsy, depression, mania, epilepsy, schizophrenia and so on
13. Uncontrolled diabetes, hypertension or thyroid disease
14. Pregnant women and lactating women or patients with pregnancy plans and not willing to use contraception during the study period
15. Participate in other clinical studies at the same time
16. Patients unsuitable for the research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
Number of participants who relapse | 96 weeks
  The total number of relapse (HBV DNA>2000 IU/ml on 2 separate occasions 1 months apart) during the research period.

SECONDARY OUTCOMES:
Number of participants who relapse | 48 weeks
  The total number of relapse (HBV DNA>2000 IU/ml on 2 separate occasions 1 months apart) during the research period.
Number of participants who achieve HBsAg seroconversion | At the point of discontinuation of PegIFN therapy
  To investigate whether Peg-IFN alfa-2a can improve the HBsAg seroconversion in CHB patients at the point of discontinuation of PegIFN therapy compared to the control group ,which will be measured by the number of participants who achieve HBsAg seroconversion. Pegasys 24 weeks Group:24 weeks and Pegasys 48 weeks Group:48 weeks
Number of participants who achieve HBsAg seroconversion | 24,48,72 weeks post-discontinuation of PegIFN therapy
  To investigate whether Peg-IFN alfa-2a can improve the HBsAg seroconversion in CHB patients at 24,48 or 72 weeks post-discontinuation of PegIFN therapy compared to the control group ,which will be measured by the number of participants who achieve HBsAg seroconversion. Pegasys 24 weeks Group:48,72,96 weeks and Pegasys 48 weeks Group:72,96 weeks
HBsAg changes from Baseline | 12,24 and 48 weeks
  Pegasys 24 weeks Group:12,24 weeks and Pegasys 48 weeks Group:12,24,48 weeks
Predictive value of other markers for recurrence after NUC withdrawal | 48 weeks and 96 weeks
  To investigate whether the other markers including HBcAb quantification and so on can predict the recurrence of hepatitis B.

CONTACTS AND LOCATIONS:
Overall Officials: Jiming Zhang, M.D., Principal Investigator — Huashan Hospital
Locations (19):
- China (19):
  - Wuhan Seventh People's Hospital, Wuhan, Hubei
  - Changzhou Third People's Hospital, Changzhou, Jiangsu
  - First Affiliated Hospital of Zhejiang University, Hangzhou, Jiangsu
  - People's Hospital of Jiangsu Province, Nanjing, Jiangsu
  - Nantong Third People's Hospital, Nantong, Jiangsu
  - Suzhou Fifth People's Hospital, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Taicang People's Hospital, Taicang, Jiangsu
  - Wuxi Infectious Disease Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu
  - Shandong Provincial Hospital, Jinan, Shandong
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Changhai Hospital Affiliated to Second Military Medical University, Shanghai
  - Huashan Hospital Affiliated to Fudan University, Shanghai
  - Ruijin Hospital Affiliate to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai Public Health Clinical Center, Shanghai
  - Shanghai Third People's Hospital, Shanghai
  - Shuguang Hospital Affiliate to Shanghai University of Traditional Chinese Medicine, Shanghai
  - The Infectious Disease Hospital of Shanghai Huangpu Distric, Shanghai

REFERENCES:
- [Result] Ganem D, Prince AM. Hepatitis B virus infection--natural history and clinical consequences. N Engl J Med. 2004 Mar 11;350(11):1118-29. doi: 10.1056/NEJMra031087. No abstract available. PMID 15014185
- [Result] Liang X, Bi S, Yang W, Wang L, Cui G, Cui F, Zhang Y, Liu J, Gong X, Chen Y, Wang F, Zheng H, Wang F, Guo J, Jia Z, Ma J, Wang H, Luo H, Li L, Jin S, Hadler SC, Wang Y. Epidemiological serosurvey of hepatitis B in China--declining HBV prevalence due to hepatitis B vaccination. Vaccine. 2009 Nov 5;27(47):6550-7. doi: 10.1016/j.vaccine.2009.08.048. Epub 2009 Sep 1. PMID 19729084
- [Result] Liang X, Bi S, Yang W, Wang L, Cui G, Cui F, Zhang Y, Liu J, Gong X, Chen Y, Wang F, Zheng H, Wang F, Guo J, Jia Z, Ma J, Wang H, Luo H, Li L, Jin S, Hadler SC, Wang Y. Evaluation of the impact of hepatitis B vaccination among children born during 1992-2005 in China. J Infect Dis. 2009 Jul 1;200(1):39-47. doi: 10.1086/599332. PMID 19469708
- [Result] Lu FM, Zhuang H. Management of hepatitis B in China. Chin Med J (Engl). 2009 Jan 5;122(1):3-4. No abstract available. PMID 19187608
- [Result] European Association For The Study Of The Liver. EASL clinical practice guidelines: Management of chronic hepatitis B virus infection. J Hepatol. 2012 Jul;57(1):167-85. doi: 10.1016/j.jhep.2012.02.010. Epub 2012 Mar 20. No abstract available. PMID 22436845
- [Result] Lok AS, McMahon BJ. Chronic hepatitis B: update 2009. Hepatology. 2009 Sep;50(3):661-2. doi: 10.1002/hep.23190. No abstract available. PMID 19714720
- [Result] Liaw YF, Leung N, Kao JH, Piratvisuth T, Gane E, Han KH, Guan R, Lau GK, Locarnini S; Chronic Hepatitis B Guideline Working Party of the Asian-Pacific Association for the Study of the Liver. Asian-Pacific consensus statement on the management of chronic hepatitis B: a 2008 update. Hepatol Int. 2008 Sep;2(3):263-83. doi: 10.1007/s12072-008-9080-3. Epub 2008 May 10. PMID 19669255
- [Result] 中华医学会肝病学分会,中华医学会感染病学分会.慢性乙型肝炎防治指南(2010年版).中华内科杂志,2011;50(2):168-179
- [Result] Kim YJ, Kim K, Hwang SH, Kim SS, Lee D, Cheong JY, Cho SW. Durability after discontinuation of nucleos(t)ide therapy in chronic HBeAg negative hepatitis patients. Clin Mol Hepatol. 2013 Sep;19(3):300-4. doi: 10.3350/cmh.2013.19.3.300. Epub 2013 Sep 30. PMID 24133668
- [Result] Liu F, Wang L, Li XY, Liu YD, Wang JB, Zhang ZH, Wang YZ. Poor durability of lamivudine effectiveness despite stringent cessation criteria: a prospective clinical study in hepatitis B e antigen-negative chronic hepatitis B patients. J Gastroenterol Hepatol. 2011 Mar;26(3):456-60. doi: 10.1111/j.1440-1746.2010.06492.x. PMID 21332542
- [Result] Seto WK, Hui AJ, Wong VW, Wong GL, Liu KS, Lai CL, Yuen MF, Chan HL. Treatment cessation of entecavir in Asian patients with hepatitis B e antigen negative chronic hepatitis B: a multicentre prospective study. Gut. 2015 Apr;64(4):667-72. doi: 10.1136/gutjnl-2014-307237. Epub 2014 May 15. PMID 24833635
- [Result] Jeng WJ, Sheen IS, Chen YC, Hsu CW, Chien RN, Chu CM, Liaw YF. Off-therapy durability of response to entecavir therapy in hepatitis B e antigen-negative chronic hepatitis B patients. Hepatology. 2013 Dec;58(6):1888-96. doi: 10.1002/hep.26549. Epub 2013 Oct 17. PMID 23744454
- [Result] Micco L, Peppa D, Loggi E, Schurich A, Jefferson L, Cursaro C, Panno AM, Bernardi M, Brander C, Bihl F, Andreone P, Maini MK. Differential boosting of innate and adaptive antiviral responses during pegylated-interferon-alpha therapy of chronic hepatitis B. J Hepatol. 2013 Feb;58(2):225-33. doi: 10.1016/j.jhep.2012.09.029. Epub 2012 Oct 6. PMID 23046671
- [Result] Chen J, Wang Y, Wu XJ, Li J, Hou FQ, Wang GQ. Pegylated interferon alpha-2b up-regulates specific CD8+ T cells in patients with chronic hepatitis B. World J Gastroenterol. 2010 Dec 28;16(48):6145-50. doi: 10.3748/wjg.v16.i48.6145. PMID 21182232
- [Result] Marcellin P, Bonino F, Yurdaydin C, Hadziyannis S, Moucari R, Kapprell HP, Rothe V, Popescu M, Brunetto MR. Hepatitis B surface antigen levels: association with 5-year response to peginterferon alfa-2a in hepatitis B e-antigen-negative patients. Hepatol Int. 2013 Mar;7(1):88-97. doi: 10.1007/s12072-012-9343-x. Epub 2012 Mar 23. PMID 23518903
- [Result] Ning Q, Han M, Sun Y, Jiang J, Tan D, Hou J, Tang H, Sheng J, Zhao M. Switching from entecavir to PegIFN alfa-2a in patients with HBeAg-positive chronic hepatitis B: a randomised open-label trial (OSST trial). J Hepatol. 2014 Oct;61(4):777-84. doi: 10.1016/j.jhep.2014.05.044. Epub 2014 Jun 7. PMID 24915612
- [Result] Ouzan D, Penaranda G, Joly H, Khiri H, Pironti A, Halfon P. Add-on peg-interferon leads to loss of HBsAg in patients with HBeAg-negative chronic hepatitis and HBV DNA fully suppressed by long-term nucleotide analogs. J Clin Virol. 2013 Dec;58(4):713-7. doi: 10.1016/j.jcv.2013.09.020. Epub 2013 Sep 29. PMID 24183313
- [Derived] Li F, Qu L, Liu Y, Wu X, Qi X, Wang J, Zhu H, Yang F, Shen Z, Guo Y, Zhang Y, Yu J, Mao R, Zhang Q, Zhang F, Chen L, Huang Y, Zhang X, Li Q, Zhang W, Zhang J. PegIFN alpha-2a reduces relapse in HBeAg-negative patients after nucleo(s)tide analogue cessation: A randomized-controlled trial. J Hepatol. 2025 Feb;82(2):211-221. doi: 10.1016/j.jhep.2024.07.019. Epub 2024 Jul 31. PMID 39094743